CLINICAL TRIAL: NCT02043665
Title: A Phase 1, Dose-finding and Signal-seeking Study of the Safety & Efficacy of Intravenous CAVATAK® Alone and in Combination With Pembrolizumab in Patients With Late Stage Solid Tumours (VLA-009 STORM / KEYNOTE-200)
Brief Title: CVA21 and Pembrolizumab in NSCLC & Bladder Cancer (VLA-009 STORM/ KEYNOTE-200)
Acronym: STORM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-200; VLA 009/ KEYNOTE-200 (Other: Viralytics Study ID); 2012-005256-42 (EudraCT Number)
Record Dates: First submitted 2014-01-19; First posted 2014-01-23 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer; Bladder Cancer
Keywords: CAVATAK; KEYNOTE-200; pembrolizumab; lung cancer; bladder cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Lung Neoplasms | interventions — pembrolizumab

ARMS (1):
- CVA21/pembrolizumab (Experimental): CVA21/pembrolizumab
  Interventions: Biological: CVA21/pembrolizumab

INTERVENTIONS:
Biological: CVA21/pembrolizumab

SUMMARY:
The purpose of this trial is to assess the ability of CVA21, either alone (Part A) or in combination with pembrolizumab (Part B), to reach and to replicate in existing tumors (while sparing normal cells) and to establish a safe multi-dose schedule of the virus for the treatment of solid tumors where enhanced expression of ICAM-1 and/ or DAF receptor occurs.

This trial consists of 2 sequential parts: VLA-009 (Part A) conducted only in the UK and employed CVA21 as a monotherapy in NSCLC, castrate-resistant prostate cancer, melanoma and bladder cancer. VLA-009 (Part B) conducted in the US, AUS and UK employs CVA21 with pembrolizumab in NSCLC and bladder cancer.

Both VLA-009A and VLA-009B are open-label, multi-center, ascending dose escalation (3+3 design) dose-finding and signal-seeking studies.

Part A of the study is now complete and closed to enrolment. Part B is currently enrolling.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed (1) NSCLC, (2) bladder cancer, (3) castrate-resistant prostate cancer which are metastatic, or (4) stage 3C or stage 4 melanoma.
* VLA009A: Locally advanced and/or metastatic disease for which curative surgery and/or radiation therapy is not possible and judged not to be a candidate for the current standard of care treatment. VLA009B: locally advanced and/or metastatic disease and judged to be a candidate for pembrolizumab to be used in combination with CVA21.
* All subjects in Cohort 3 or Phase 2 dose (P2D) must have a lesion accessible for FNA or core or open biopsy on day 8 of the first treatment cycle.
* No CVA21 neutralising antibody (≤ 1:16)
* Measurable or evaluable disease

Exclusion Criteria:

* Second primary malignancy within the past 2 years (except non-melanoma skin cancer, in situ carcinoma of the cervix, breast cancer)
* Concurrent immunosuppressive therapy and no known immunosuppressive disease other than primary tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Response rate assessed according to immune-related RECIST 1.1 criteria | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hardev Pandha, MD, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (18):
- United States (9):
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Miami, Coral Gables, Florida
  - Advocate Health, Niles, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (6):
  - Tasman Oncology Research, Southport, Queensland
  - Monash Health, Clayton, Victoria
  - St Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Epworth HealthCare, Richmond, Victoria
  - St John of God Healthcare, Subiaco, Western Australia
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust, Chelsea
  - Royal Surrey County Hospital, Guildford
  - St. James University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rudin CM, Pandha HS, Zibelman M, Akerley WL, Harrington KJ, Day D, Hill AG, O'Day SJ, Clay TD, Wright GM, Jennens RR, Gerber DE, Rosenberg JE, Ralph C, Campbell DC, Curti BD, Merchan JR, Ren Y, Schmidt EV, Guttman L, Gupta S. Phase 1, open-label, dose-escalation study on the safety, pharmacokinetics, and preliminary efficacy of intravenous Coxsackievirus A21 (V937), with or without pembrolizumab, in patients with advanced solid tumors. J Immunother Cancer. 2023 Jan;11(1):e005007. doi: 10.1136/jitc-2022-005007. PMID 36669791